CLINICAL TRIAL: NCT05659537
Title: A 24-week Multicenter, Open-label, Single-arm Study to Evaluate Safety in Patients With Type 2 Diabetes Mellitus in India Treated With Dulaglutide
Brief Title: A Study of Dulaglutide (LY2189265) in Participants With Type 2 Diabetes Mellitus in India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18550; H9X-IN-GBGR (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-12-15; First posted 2022-12-21 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Adult; GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dulaglutide (Experimental): * Participants received once-weekly (QW) subcutaneous (SC) dulaglutide injections for 24 weeks, starting with either 1.5 milligrams (mg) as combination therapy or 0.75 mg as combination therapy or monotherapy (at the discretion of the investigator).
  * For participants reporting gastrointestinal adverse events (GI AEs) after starting the 1.5 mg dulaglutide dose, the investigator reduced the dose to 0.75 mg for 2 to 3 weeks. Thereafter, the 1.5 mg dose was reintroduced.
  Interventions: Drug: Dulaglutide

INTERVENTIONS:
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265

SUMMARY:
The main purpose of this study is to evaluate safety of dulaglutide in participants with type 2 diabetes mellitus in India.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of type 2 diabetes mellitus (T2DM) of at least 1-year duration currently treated with stable doses of oral antihyperglycemic medications with or without stable doses of basal or premix insulin for the last 3 months prior to screening
* Have hemoglobin A1c (HbA1c) greater than or equal to (≥) 7.5 percent (%) and less than or equal to (≤) 11.5%, both inclusive, at screening
* Have body mass index (BMI) ≥ 23 kilogram/square meter (kg/m²)

Exclusion Criteria:

* A diagnosis of type 1 diabetes mellitus (T1DM) or latent autoimmune diabetes, or specific type of diabetes other than T2DM
* Been treated with antihyperglycemic medication like glucagon-like peptide receptor agonists (GLP-1 RA) or have a prior history of any contraindication to GLP-1 RA therapy within 3 months prior to screening or estimated glomerular filtration rate (eGFR) <15 milliliter/minute (ml/min)/1.73 square meter (m²)
* Participants have known hypersensitivity or allergy to dulaglutide or its excipients
* Participants are on systemic steroids for any period of more than 14 days
* Participants have severe gastrointestinal (GI) disease, including severe gastroparesis
* Participants have an active or untreated malignancy, except for successfully treated basal or squamous cell carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- India (7):
  - Medlink Hospital Opp Someshwara Jain Temple, Ahmedabad, Ambavadi
  - Life Care Hospital and Research Centre, Bangalore, Karnataka
  - Grant Medical Foundation - Ruby Hall Clinic, Pune, Maharashtra
  - Akshay Hospital, Pune, Maharashtra
  - Lifepoint Multispecialty Hsptl, Wakad, Pune
  - Kovai Diabetes Speciality Center and Hospital, Coimbatore, Tamil Nadu
  - Virinchi Hospital, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dulaglutide
Started | 212
Received at Least One Dose of Dulaglutide (Safety Population) | 200 (Received at least one dose of 1.5 mg and 0.75 mg dulaglutide = 165; received at least one dose of 1.5 mg dulaglutide only = 21 and received at least one dose of 0.75 mg dulaglutide only = 14.)
Received at Least One Dulaglutide Dose and Had at Least One HbA1c Measurement Post-study Treatment | 189
Completed | 185
Not Completed | 27
Not completed — Adverse Event | 5
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 13
Not completed — Migration from the Study Site Such That Follow Up Visits are not Possible | 3
Not completed — Participant had low absolute neutrophil count value | 1
Not completed — Participant was suffering from anaemia | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dulaglutide dose and had at least one HbA1c measurement post-study treatment.
Groups:
- Dulaglutide: * Participants received QW dulaglutide SC injections for 24 weeks, starting with either 1.5 mg as combination therapy or 0.75 mg as combination therapy or monotherapy (at the discretion of the investigator).
  * For participants reporting GI AEs after starting the 1.5 mg dulaglutide dose, the investigator reduced the dose to 0.75 mg for 2 to 3 weeks. Thereafter, the 1.5 mg dose was reintroduced.
Arm/Group | Dulaglutide
Number analyzed (Participants) | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (10.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 189
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 189
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  India | 189

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Adverse Events (AEs) - Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Deaths
Description: * An AE was any untoward medical occurrence in a participant who was administered an investigational product that did not necessarily have a causal relationship with the treatment. A TEAE was defined as an AE that occurred post-dose or was present prior to dosing and became more severe post-dose.
  * An SAE was any AE from the study that resulted in one of the following: death, initial or prolonged inpatient hospitalization, a life-threatening experience (i.e., immediate risk of dying), persistent or significant disability/incapacity, congenital anomaly/birth defect, or important medical events that might not have been immediately life-threatening or resulted in death or hospitalization but might have jeopardized the participant or required intervention to prevent one of the other outcomes listed in the definition above.
  * A summary of SAEs and other non-serious AEs, regardless of causality, is located in the reported Adverse Events section of this record.
Time Frame: Baseline through Follow-up (up to 28 weeks)
Population: All participants who received at least one dulaglutide dose and had at least one HbA1c measurement post-study treatment. As prespecified in the statistical analysis plan, the primary and secondary outcomes were planned to be analyzed and reported by dose level only if the proportion in each arm was more than 20 percent (%). However, the percentage in the 1.5 mg only or 0.75 mg only dulaglutide arm was lower than 20 %. Hence, outcomes are reported for the overall dulaglutide treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Dulaglutide
Number analyzed (Participants) | 189
Participants
  TEAEs | 106
  SAEs | 1
  Deaths | 0

2. Primary Outcome: Number of Participants With One or More Hypoglycemic Events, Including Severe Hypoglycemic Events.
Description: Hypoglycemia events were defined as those with blood glucose (BG) levels less than (<) 70 milligrams per deciliter (mg/dL). Severe hypoglycemia events were defined as those with severe cognitive impairment requiring the assistance of another person to actively administer carbohydrates, glucagon, or other resuscitative actions. These events could be associated with sufficient neuroglycopenia to induce seizures or coma. The total number of participants who experienced hypoglycemia events, including severe hypoglycemia, was summarized cumulatively.
Time Frame: Baseline through Follow-up (up to 28 weeks)
Population: All participants who received at least one dulaglutide dose and had at least one HbA1c measurement post-study treatment. As prespecified in the statistical analysis plan, the primary and secondary outcomes were planned to be analyzed and reported by dose level only if the proportion in each arm was more than 20%. However, the percentage in the 1.5 mg only or 0.75 mg only dulaglutide arm was lower than 20%. Hence, outcomes are reported for the overall dulaglutide treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Dulaglutide
Number analyzed (Participants) | 189
Participants | 13

3. Primary Outcome: Percentage of Participants Reporting AEs and SAEs From Baseline to Week 24
Description: The percentage of participants who reported AEs and SAEs was calculated by dividing the total number of affected participants by the number of participants analyzed, then multiplying by 100. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the reported Adverse Events section of this record.
Time Frame: Baseline through Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Dulaglutide
Number analyzed (Participants) | 189
percentage of participants
  AEs | 51.9
  SAEs | 0.5

4. Primary Outcome: Number of Participants With One or More Gastrointestinal (GI) AEs From Baseline to Week 24
Description: The number of participants who experienced at least one or more GI AEs of nausea, vomiting, and diarrhoea were summarized cumulatively. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the reported Adverse Events section of this record.
Time Frame: Baseline through Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dulaglutide
Number analyzed (Participants) | 189
Participants | 48

5. Secondary Outcome: Mean Change in HbA1c From Baseline to Week 24
Description: HbA1c is the glycosylated fraction of hemoglobin A. It is measured to identify average plasma glucose concentration over prolonged periods of time. The mean change in HbA1c levels was calculated using descriptive analysis, with baseline HbA1c as a covariate. Missing endpoints were addressed using the last observation carried forward (LOCF) method.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Dulaglutide
Number analyzed (Participants) | 189
Percentage of HbA1c | -1.41 (1.422)

ADVERSE EVENTS:
Time Frame: From baseline until safety follow-up (up to 28 weeks)
Description: All participants who had received at least one dose of dulaglutide.
Groups:
- 1.5 mg/0.75 mg Dulaglutide (Both Doses): Participants in this arm received SC injections of both 1.5 mg and 0.75 mg dulaglutide QW doses at different points during the 24-week treatment period.
- 1.5 mg Dulaglutide Only: Participants in this arm received SC injections of only 1.5 mg of dulaglutide QW over a 24-week treatment period.
- 0.75 mg Dulaglutide Only: Participants in this arm received SC injections of only 0.75 mg of dulaglutide QW over a 24-week treatment period.
Arm/Group | 1.5 mg/0.75 mg Dulaglutide (Both Doses) | 1.5 mg Dulaglutide Only | 0.75 mg Dulaglutide Only
All-Cause Mortality (participants affected / at risk) | 0/165 | 0/21 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/165 | 0/21 | 0/14
Other Adverse Events (participants affected / at risk) | 100/165 | 8/21 | 6/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.5 mg/0.75 mg Dulaglutide (Both Doses) (N=165) | 1.5 mg Dulaglutide Only (N=21) | 0.75 mg Dulaglutide Only (N=14)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.5 mg/0.75 mg Dulaglutide (Both Doses) (N=165) | 1.5 mg Dulaglutide Only (N=21) | 0.75 mg Dulaglutide Only (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 17 (17) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 6 (8) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 13 (17) | 3 (4) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 23 (23) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 25 (25) | 1 (1) | 1 (1)
Asthenia (General disorders) | 4 (4) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Albumin urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 4 (4) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 11 (11) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 9 (9) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypolipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 9 (9) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-06-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT05659537/Prot_002.pdf
  • Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT05659537/SAP_001.pdf